CLINICAL TRIAL: NCT01312506
Title: Procurement of Central Nervous System and Extracranial Tumor Tissues, Cerebrospinal Fluid, and Serum/Plasma From Patients With Metastatic Melanoma to the CNS and Respective Controls for Gene Expression and Proteomic Profiling
Brief Title: Collection of Cerebrospinal Fluid and Tumor Tissue in Subjects With Metastatic Melanoma and Controls
Status: Withdrawn | Type: Observational
Why Stopped: Trial experienced funding issues, was never opened to accrual.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 10-067
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Melanoma; CNS Metastases
Keywords: metastatic; melanoma; CNS
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Subjects undergoing a craniotomy: This group will include those subjects who have consented to have either a craniotomy or a laminectomy to resect an intramedullary tumor.
- Metastases, no craniotomy: These subjects have metastases but have either chosen not to undergo removal of the cancer or their neurosurgeon does not recommend surgical approach or they have been diagnosed with metastatic melanoma but do not have CNS metastases.
- Healthy Volunteers: Subjects who do not have known melanoma or metastases.

SUMMARY:
This study has two ultimate goals:

1. Understand how the original melanoma from the skin spreads to the CNS. In order to study this we need to collect (and compare) the original skin melanoma, the CNS melanoma, as well as any other melanoma that has not metastasized to the CNS.
2. Develop a diagnostic blood test that will early identify subjects at high risk for developing CNS metastasis or patients who may already have CNS metastasis but the MRI or the CAT scan cannot yet detect it. Thus, the investigators plan to collect CSF from subjects like you who have melanoma CNS metastases in order to confirm the presence of this biomarker.

ELIGIBILITY:
Inclusion Criteria:

1. Regarding patients with distant metastatic melanoma and established melanoma CNS metastases who are scheduled for craniotomy:

   * Histologically confirmed, primary cutaneous melanoma, metastatic to the CNS (brain OR spinal cord OR carcinomatous meningitis) based on:

     * Pathologic confirmation (i.e. prior craniotomy) OR
     * Radiography (brain MRI or CT scan with intravenous contrast)
   * Patients must have no contraindications for and be able to undergo lumbar puncture for CSF collection
   * Hemoglobin level of 8g/dL or higher. This can be drawn on the day of consent, or will be acceptable if documented from a previous visit within the prior 30 days
   * Subjects must have provided written, informed consent (ICF) prior to any study procedures
   * Subjects must provide a FFPE tissue block containing a biopsy from the primary site
2. Regarding patients with distant metastatic melanoma and established melanoma CNS metastases who are not having a craniotomy and before they undergo external beam irradiation or stereotactic radiosurgery (patient's and/or neurosurgeon's preference):

   * Histologically confirmed melanoma (unknown primary, mucosal, ocular are allowed), metastatic to the CNS (brain OR spinal cord OR carcinomatous meningitis) based on

     * Pathologic confirmation (i.e. prior craniotomy) and/or
     * Radiography (brain MRI or CT scan with intravenous contrast)
   * Patients must have no contraindications for and be able to undergo lumbar puncture for CSF collection
   * Hemoglobin level of 8g/dL or higher. This can be drawn on the day of consent, or will be acceptable if documented from a previous visit within the prior 30 days
   * Subjects must have provided written ICF prior to any study procedures
3. Regarding patients who have distant metastatic melanoma without radiographically detectable melanoma CNS metastases but are willing to undergo lumbar puncture:

   * Histologically confirmed melanoma (unknown primary, mucosal, ocular are allowed),
   * Patients must have no contraindications to lumbar puncture
   * Hemoglobin level of 8g/dL or higher. This can be drawn on the day of consent, or will be acceptable, if documented from a previous visit within the prior 30 days
   * Subjects must have provided written ICF prior to any study procedures
4. Regarding healthy volunteers

   * Patients must have no contraindications to lumbar puncture (see Table 1)
   * Patient must answer NO to all questions listed in Appendix B
   * Hemoglobin level of 8g/dL or higher. This can be drawn on the day of consent or will be acceptable if documented from a previous visit within the prior 30 days
   * Subjects must have provided written, ICF prior to any study procedures

Exclusion Criteria:

* For study subjects, patients with extradural lesions, i.e. those that originate from the bone (calvarium or vertebrae), will not be considered.
* Any significant psychiatric disease, medical intervention, or other conditions, which in the opinion of the Investigators, could impair proper discussion of the informed consent or compromise participation to the clinical trial.
* Active systemic treatment for metastatic melanoma within 2 days from the collection of specimens (brain tumor tissue, peripheral blood, CSF). Corticosteroids, other immunosuppressive anti-inflammatory and anti-epileptic medications are allowed.
* Patients who have undergone whole brain irradiation therapy within the last 30 days. Therefore neither CNS lesions nor CSF are considered suitable for collection.
* Patients with growing CNS lesions at an area that has previously undergone radiosurgery within 3 months prior to enrollment in this study. Therefore CNS tumors from previously irradiated areas using radiosurgery are not considered suitable for collection although CSF is allowed for collection.
* Brain abscess.
* Patients with new focal findings on neurological examination.
* Infected skin over the lumbar puncture needle entry site.
* Other conditions that at the opinion of the investigator are contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Moschos, MD, Principal Investigator — University of Pittsburgh